CLINICAL TRIAL: NCT04772365
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Administered SHR-1819 in Healthy Subjects
Brief Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Dose Escalation Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1819-101
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2021-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1819
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1819 — SHR-1819 will be subcutaneously administered with different dose levels;
  Arms: Treatment group A
Drug: Placebo — Placebo will be subcutaneously administered with different dose levels;
  Arms: Treatment group B

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, single and multiple dose escalation phase 1 study. The objective of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of subcutaneous administered SHR-1819 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial, and provides written informed consent.
2. Be able to comply with all the requirements and able to complete the study.
3. Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
4. No clinically significant abnormalities in medical history, general physical examination, vital signs, and laboratory tests.
5. Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods and have no plan to have a child from signing the consent form to 16 weeks after IP administration.

Exclusion Criteria:

1. Positive hepatitis B virus (HBsAg), hepatitis C virus (HCV-Ab), human immunodeficiency virus (HIV-Ab), or QuantiFERON-TB Gold tests at screening;
2. Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening (according to the date of signed consent form), or in the follow-up period of a clinical study
3. Severe injuries or surgeries within 6 months before screening or plan to do surgeries during the trial
4. Any other circumstances that, in the investigator's judgment, may increase the risk associated with the subject's participation in and completion of the study or could preclude the evaluation of the subject's response

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study（about 13 weeks）
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (about 13 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1819 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 13 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1819 administration
Pharmacokinetics-Tmax | Up to 13 weeks
  Time to Cmax of SHR-1819
Pharmacokinetics-Cmax | Up to 13 weeks
  Maximum observed concentration of SHR-1819
Pharmacokinetics-CL/F | Up to 13 weeks
  Apparent clearance of SHR-1819
Pharmacokinetics-Vz/F | Up to 13 weeks
  Apparent volume of distribution during terminal phase of SHR-1819
Pharmacokinetics-t1/2 | Up to 13 weeks
  Terminal elimination half-life of SHR-1819
Change from baseline to end of treatment for Thymus and activation-regulated chemokine（TARC/CCL17） | Up to 13 weeks
  Thymus and activation-regulated chemokine（TARC/CCL17）
Change from baseline to end of treatment for IgE | Up to 13 weeks
  IgE
Immunogenicy of SHR-1819 after administration | Up to 13 weeks]
  Anti-drug antibody
Pharmacokinetics-AUCtau for multi-dose | Start of Treatment to end of study (about 13 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1819 administration
Pharmacokinetics- Ctrough for multi-dose | Up to 13 weeks
  Minimum observed concentration of SHR-1819
Pharmacokinetics- Racc for multi-dose | Up to 13 weeks
  Accumulation ratio of SHR-1819

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Changsha, China